CLINICAL TRIAL: NCT03515525
Title: Retrospective Review of Patient Records for Analysis of Postoperative Bleeding Following Breast Surgery
Brief Title: Analysis of Hematoma Following Breast Surgery
Status: Completed | Type: Observational
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Dr. Alexandra Anker, Plastic surgery resident, University of Regensburg
Other Study IDs: 18-955-104
Record Dates: First submitted 2018-04-22; First posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Hematoma; Postoperative Bleeding
Keywords: Breast surgery; Closed-suction drains
MeSH Terms: conditions — Hematoma; Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hematoma side: Drain secretion volume prior to revision surgery on the breast side affected by hematoma.
  Interventions: Diagnostic Test: Closed-suction drain fluid volume
- Non-hematoma side: Drain secretion volume prior to revision surgery on the breast side not affected by hematoma.
  Interventions: Diagnostic Test: Closed-suction drain fluid volume

INTERVENTIONS:
Diagnostic Test: Closed-suction drain fluid volume — To evaluate the clinical value of postoperative drain fluid volume for detection of hematoma, an intra-individual comparison of drain secretion volumes between sides affected by hematoma and the uneventful contralateral breasts was performed.

SUMMARY:
A retrospective review of patients who developed hematoma following breast surgery from 2003 to 2018 in a single institution was performed. The study investigated the value of closed-suction drains regarding the quantity and quality of fluid secretion for the prediction of subcutaneous hematoma in patients undergoing breast surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who developed hematoma requiring revision following bilateral breast surgery including augmentation mammoplasty, subcutaneous mastectomy and breast reduction.

Exclusion Criteria:

* Patients who developed hematoma requiring revision following unilateral breast surgery.
* Breast surgery in absence of hematoma.
* Patients with known coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enrolled 20 subjects who developed unilateral hematoma requiring evacuation following bilateral breast surgery between January 2008 and January 2018 at our institution. Gender, age, breast surgery subtype, preoperative and postoperative hemoglobin values as well as perioperative heparinization were recorded.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-22 (Actual)

PRIMARY OUTCOMES:
Drain fluid volume | 24 hours postoperatively
  The drain fluid volume in the breast affected by hematoma was compared to the non-hematoma side.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic Surgery, University Hospital of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No